CLINICAL TRIAL: NCT01451619
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Parallel Group Study to Assess the Pharmacodynamics of MK-0524 in Subjects With Moderate to Severe Erythematotelangiectatic Rosacea. (Protocol No. 155)
Brief Title: A Study of Laropiprant (MK-0524) in Participants With Moderate to Severe Erythematotelangiectatic Rosacea (MK-0524-155)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524-155
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — MK-0524

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laropiprant (Experimental)
  Interventions: Drug: Laropiprant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo for Laropiprant

INTERVENTIONS:
Drug: Laropiprant — One 100-mg tablet orally once daily for 4 weeks
  Other Names: MK-0524
  Arms: Laropiprant
Drug: Placebo for Laropiprant — One tablet orally once daily for 4 weeks
  Arms: Placebo

SUMMARY:
This study will assess the effect of MK-0524 relative to placebo, on signs and symptoms of rosacea and to determine the safety and tolerability profile of MK-0524 in participants with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe erythematotelangiectatic rosacea with moderate to severe erythema of facial lesion
* Generally healthy excluding rosacea
* Presence of telangiectasia
* Five or less facial inflammatory lesions
* Able to restrict diet in order to avoid foods/drinks (including alcohol) that are known to exacerbate the signs/symptoms of rosacea
* Females of childbearing potential must have negative serum pregnancy test and agree to use one form of contraception

Exclusion Criteria:

* Diagnosis of skin disorders, including psoriasis, acne vulgaris, perioral dermatitis or atopic dermatitis that would interfere with the clinical evaluations of rosacea
* Using and unable to discontinue use of phosphodiesterase (PDE) 4 inhibitors, theophylline, niacin greater than 500 mg/day
* Known or suspected excessive alcohol intake
* Sensitivity to tetracyclines
* Ocular rosacea and/or blepharitis/meibomianitis
* Pregnant or breastfeeding
* Perimenopausal and has symptoms that cause flushing that may affect rosacea
* Initiated hormonal method of birth contraception within 4 months of baseline, discontinues use during the course of the study, or changes hormonal method within 4 months
* Active mycobacterial infection of any species within 3 years
* History of mycobacterium tuberculosis infection
* History of recurrent bacterial infection
* Congenital or acquired immunodeficiency common variable immunodeficiency (CVID), Hepatitis B surface antigen positive or Hepatitis B core antibody positive
* Human immunodeficiency virus (HIV) infection
* Positive for hepatitis C antibodies
* Malignancy or has had a history of malignancy greater than 3 years prior
* Will continue to use any of the following treatments during the study: Systemic retinoids, therapeutic vitamin A supplements of greater than 10,000 units/day, systemic steroids, systemic antibiotics known to have an impact on the severity of facial rosacea, systemic treatment for acne, topical steroids, topical retinoids, topical acne treatments including prescription and over-the-counter (OTC) preparations, topical anti-inflammatory agents, topical antibiotics, topical imidazole antimycotics, cryodestruction or chemodestruction, dermabrasion, photodynamic therapy, acne surgery, intralesional steroids, X-ray therapy, pulse-dye laser, intense pulse light, astringents, abrasives, benzoyl peroxide products, sulfur containing washes, eye washes, Beta blockers, vasodilators, vasoconstrictors and/or chronic use (>14 days) of topical or systemic anti-inflammatory agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in Clinician's Erythema Assessment (CEA) Scale Score from Baseline | Baseline and Week 4

SECONDARY OUTCOMES:
Change in Patient Self Assessment (PSA) Score from Baseline | Baseline and Week 4

REFERENCES:
- [Result] Krishna R, Guo Y, Schulz V, Cord-Cruz E, Smith S, Hair S, Nahm WK, Draelos ZD. Non-obligatory role of prostaglandin D2 receptor subtype 1 in rosacea: laropiprant in comparison to a placebo did not alleviate the symptoms of erythematoelangiectaic rosacea. J Clin Pharmacol. 2015 Feb;55(2):137-43. doi: 10.1002/jcph.383. Epub 2014 Sep 4. PMID 25142778